CLINICAL TRIAL: NCT02591966
Title: Genetic Alteration After Systemic Treatment in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, MD, PhD, Division of Hematology-Oncology, Samsung Medical Center
Other Study IDs: 2014-11-015
Record Dates: First submitted 2015-10-26; First posted 2015-10-30 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood sample : whole blood
  2. Tissue : Fresh tissue, Fixed tissue (5ea of 5-10µm unstained sections),
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker group: 1. The patients who receive neoadjuvant systemic treatments:
  2. The patients who have distant metastatic sites at first and recur from surgery:
  3. The patients who are going to receive first-line chemotherapy:

SUMMARY:
The purpose of this study is to investigate effects of systemic treatments on genomic profiles in patients with breast cancer and to compare genomic profiling between premenopausal and postmenopausal women by systemic treatments in breast cancer.

DETAILED DESCRIPTION:
Prospective single arm trial using three patients' cohorts. One-hundred patients for each cohort and a total of 300 patients (600 biopsy samples) will be entered to this trial.

The hypothesis is that genomic alterations measured by CancerSCAN and cfDNA, Whole exome sequencing (WES), Whole transcriptome sequencing (WTS), FACS(Fluorescence-Activated Cell Sorting), cytokine and immunologic signature analysis would be different between pre- and post-menopausal women and would be predictive biomarkers for each cohort according to pre- and post-menopausal status. Three groups of patients will be recruited:

1. The patients who receive neoadjuvant systemic treatments:
2. The patients who have distant metastatic sites at first and recur from surgery:
3. The patients who are going to receive first-line chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 20 years
2. Patients with histologically confirmed breast cancer at three disease status

   * Patients who are going to receive neoadjuvant chemotherapy with feasible biopsy site.
   * Patients who recur from curative surgery and have distant metastasis with feasible biopsy site. ; Patients must have received adjuvant chemotherapy after curative surgery.
   * Patients who are going to first-line palliative chemotherapy with feasible biopsy site.
3. Patients with PS ECOG 0 - 2
4. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
5. Written informed consent form
6. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to study as defined below:

   * Haemoglobin ≥9.0 g/L (transfusion allowed)
   * White blood cells (WBC) > 3 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN

Exclusion Criteria:

1. Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical condition that would interfere with the subject's safety.
2. Double primary cancer (except for any cancer in remission for > 5 years, cervix cancer in situ, basal cell cancer in situ, any in situ cancers that are resected)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The patients who receive neoadjuvant systemic treatments:
  2. The patients who have distant metastatic sites at first and recur from surgery:
  3. The patients who are going to receive first-line chemotherapy:
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Genomic profiling will be assessed by tissue sampling and blood. | 2year
  Tissue and blood will be tested for CancerSCAN, cfDNA, WES, WTS, FACS, cytokine and immunologic signature analysis platform.NAC to study the multiscale relationships among DCE-MRI features, NGS data, and pathologic response to NAC and to evaluate the role of radiogenomics in predicting pathologic response of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea